CLINICAL TRIAL: NCT02823964
Title: An Open-Label Study Evaluating the Efficacy and Safety of Liprotamase in Subjects With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis
Brief Title: EASY: Extended Access to Sollpura Over Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN-EPI3334
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Exocrine Pancreatic Insufficiency; Cystic Fibrosis
Keywords: exocrine pancreatic insufficiency; cystic fibrosis; pancreatic enzyme replacement therapy
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis | interventions — liprotamase lipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liprotamase (Experimental): Oral, soluble, non-enterically coated, non-porcine, pancreatic enzyme replacement
  Interventions: Drug: Liprotamase

INTERVENTIONS:
Drug: Liprotamase — Oral, soluble, non-enterically coated, non-porcine, pancreatic enzyme replacement
  Other Names: Sollpura

SUMMARY:
Liprotamase consists of 3 soluble, non-porcine digestive enzymes, lipase, protease, and amylase, combined in a fixed ratio. Liprotamase is stable in the stomach and can be formulated without enteric coating for administration either as a capsule or as a dosing solution dissolved in water or juice.

DETAILED DESCRIPTION:
The purpose of the present study is to evaluate the safety of long-term use of liprotamase in the management of cystic fibrosis-related exocrine pancreatic insufficiency

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with cystic fibrosis-related exocrine pancreatic insufficiency who received liprotamase and completed Study AN-EPI3331 (SOLUTION: Study of Oral Liprotamase Unit-Matched Therapy Of Non-Porcine Origin in Patients With Cystic Fibrosis)

Exclusion Criteria:

* Any medical, psychological, or social condition that may put the subject at increased risk by participating in this study.
* Females who are nursing, pregnant, intending to become pregnant, or intending to nurse during the time of the study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (3):
  - Investigator Site 114, Aurora, Colorado
  - Investigator Site 134, Jackson, Mississippi
  - Investigator Site 121, Burlington, Vermont
- Investigator Site 501, Brno, Czechia
- Hungary (4):
  - Investigator Site 303, Debrecen, Hajdú-Bihar
  - Investigator Site 302, Törökbálint, Pest County
  - Investigator Site 304, Mosdós, Somogy County
  - Investigator Site 301, Ajka, Veszprém megye
- Investigator Site 601, Jerusalem, Israel
- Poland (5):
  - Investigator Site 203, Karpacz
  - Investigator Site 206, Lodz
  - Investigator Site 205, Lublin
  - Investigator Site 202, Rabka-Zdrój
  - Investigator Site 209, Rzeszów
- Investigator Site 401, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liprotamase
Started | 25
Completed | 20
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Liprotamase
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.94 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety, as Measured by Number of Participants With Adverse Events Including Clinical or Laboratory Abnormalities
Description: Descriptive analysis
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Liprotamase
Number analyzed (Participants) | 25
Participants
  Safety population | 25
  total number of subjects with adverse events | 9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Liprotamase
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liprotamase (N=25)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 (2)
Scalded Skin (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liprotamase (N=25)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hemoptoe (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infective pulmonary exacerbation of CF (Infections and infestations) | 4 (4)
Viral infection (Infections and infestations) | 2 (2)
Scalded skin (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2)
Kidney stone (Renal and urinary disorders) | 2 (2)
Investigations (Investigations) | 3 (3)
Minocycline allergy (Immune system disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT02823964/Prot_SAP_000.pdf